CLINICAL TRIAL: NCT01807858
Title: The Effects of Synbiotics on Morbidity and Mortality in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, Assoc Prof, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 68/16.Oct.2012
Record Dates: First submitted 2012-12-24; First posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Necrotizing Enterocolitis; Sepsis
Keywords: Necrotizing enterocolitis; Sepsis; Length of hospital stay; Mortality
MeSH Terms: conditions — Enterocolitis, Necrotizing; Sepsis | interventions — maltodextrin; Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bifidobacterium lactis (Active Comparator): 5 billion Bifidobacterium lactis
  Interventions: Dietary Supplement: Bifidobacterium lactis plus İnülin; Other: Maltodextrin; Dietary Supplement: İnulin
- İnulin (Active Comparator): 900 mg İnulin per day will be given
  Interventions: Dietary Supplement: Bifidobacterium lactis; Dietary Supplement: Bifidobacterium lactis plus İnülin; Other: Maltodextrin
- Maltodextrin (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Bifidobacterium lactis; Dietary Supplement: Bifidobacterium lactis plus İnülin; Dietary Supplement: İnulin
- Bifidobacterium lactis plus İnülin (Active Comparator): 5 billion active Bifidobacterium lactis plus 900 mg İnülin per day
  Interventions: Dietary Supplement: Bifidobacterium lactis; Other: Maltodextrin; Dietary Supplement: İnulin

INTERVENTIONS:
Dietary Supplement: Bifidobacterium lactis — 5 billion active Bifidobacterium lactis
  Arms: Bifidobacterium lactis plus İnülin; Maltodextrin; İnulin
Dietary Supplement: Bifidobacterium lactis plus İnülin — 5 billion Bifidobacterium lactis plus 900 mg İnülin per day will be given
  Other Names: 5 billion Bifidobacterium lactis plus 900 mg İnülin
  Arms: Bifidobacterium lactis; Maltodextrin; İnulin
Other: Maltodextrin — Maltodextrin
  Arms: Bifidobacterium lactis; Bifidobacterium lactis plus İnülin; İnulin
Dietary Supplement: İnulin — 900 mg inulin per day will be given
  Arms: Bifidobacterium lactis; Bifidobacterium lactis plus İnülin; Maltodextrin

SUMMARY:
Study, the inclusion of very low birth weight premature infants followed in Dr.Sami Ulus Maternity and Children Training and Research Hospital, Department of Neonatology; be randomized to very low birth weight premature infants began eating until you are discharged from the hospital once a day to feed a group+ 900 mg of 5 billion active Bifidobacterium lactis, the addition of chicory inulin, in the other group given placebo; Patients taking weekly blood cultures, the presence of residues in both groups during feeding, to evaluate the incidence of NEC and sepsis are planned. Randomization and the number of patients planned to separate into groups.

DETAILED DESCRIPTION:
Patients separated into four groups using the sealed envelope method.

ELIGIBILITY:
Inclusion Criteria:

* VLBW infants admitted to NICU at the first 7 days of life

Exclusion Criteria:

* expected life lower than 7 days,
* babies who could not be fed (any metabolic disorders, gastrointestinal system surgical disorders etc.),
* severe asphyxia,
* severe congenital anomaly

Max Age: 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Necrotizing enterocolitis | 8 weeks
  Developing of >= grade 2 necrotizing enterocolitis suggested by radiological investigation

SECONDARY OUTCOMES:
length of hospital stay | 16 weeks
  length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Dilli, MD, Principal Investigator — Assoc Prof
Locations (4):
- Turkey (Türkiye) (4):
  - Şevket Yılmaz Research Hospital, Bursa
  - Diyarbakır Research Hospital, Diyarbakır
  - Okmeydani Research Hospital, Istanbul
  - Umraniye Research Hospital, Istanbul

REFERENCES:
- [Background] Fouhy F, Ross RP, Fitzgerald GF, Stanton C, Cotter PD. Composition of the early intestinal microbiota: knowledge, knowledge gaps and the use of high-throughput sequencing to address these gaps. Gut Microbes. 2012 May-Jun;3(3):203-20. doi: 10.4161/gmic.20169. Epub 2012 May 1. PMID 22572829
- [Derived] Dilli D, Aydin B, Fettah ND, Ozyazici E, Beken S, Zenciroglu A, Okumus N, Ozyurt BM, Ipek MS, Akdag A, Turan O, Bozdag S. The propre-save study: effects of probiotics and prebiotics alone or combined on necrotizing enterocolitis in very low birth weight infants. J Pediatr. 2015 Mar;166(3):545-51.e1. doi: 10.1016/j.jpeds.2014.12.004. Epub 2015 Jan 13. PMID 25596096
- See also: Are Probiotics Safe For Newborns? | LIVESTRONG.COM — http://www.livestrong.com/article/468506-are-probiotics-safe-for-newborns/